CLINICAL TRIAL: NCT03078374
Title: A Safety and Feasibility Study of Low-intensity Anticoagulation With HeartMate 3 LVAS: A Single Center Prospective Controlled Study (MAGENTUM 1)
Brief Title: MAGENTUM 1 HeartMate 3 LVAS: A Single Center Prospective Controlled Study (MAGENTUM 1)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Prof. Ivan Netuka, MD, Ph.D., Vice Chairman of Cardiac Centre, Institute for Clinical and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 2.0
Record Dates: First submitted 2017-03-02; First posted 2017-03-13 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure; Cardiovascular Diseases
Keywords: Reduced anti-coagulation, mechanical circulatory support.
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced Anticoagulation (Other): Reduced anticoagulation
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Reduced dosage to obtain lower INR range

SUMMARY:
The purpose of this study is to obtain single-center safety and feasibility data on patients managed with reduced anti-coagulation, and the incidence of thrombotic and bleeding adverse events associated with the HeartMate 3 LVAS therapy.

DETAILED DESCRIPTION:
Patients with implanted HeartMate 3 device will be bridged with heparin until target International Normalized Ratio (INR) of 2,0 - 3,0 will be reached on anticoagulation therapy with Warfarin. Along with Warfarin, Acetylsalicylic Acid (ASA) will be administered in dose of 100mg per day. Enrollment for the study will take place in 1-6 weeks post implant of HeartMate 3. Low-intensity anticoagulation protocol will be started at 6 weeks after implant. Target INR of 1,5-1,9 will be maintained and ASA will be administered in dose of 100mg per day with adjustments based on VerifyNow testing. Follow up will last for 12 months after HeartMate 3 implantation. Subsequently, the objectives of the study will be analyzed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients implanted with HeartMate 3 LVAS irrespective of an indication
* data collection for major thrombophilic mutations including anti-phospholipid syndrome and lupus anticoagulant testing prior to low-intensity protocol anticoagulation initiation has been performed
* patient will be compliant with an anticoagulation management in a judgment of the investigator
* patient in stable condition with anticipated home discharge

Exclusion Criteria:

* absence of an informed consent
* presence of additional MCS e.g. ECMO, RVAD in less than 7 days prior to low- intensity protocol anticoagulation initiation
* known history of major thrombotic event e.g. DVT
* presence of other than biological valve prosthesis in aortic position
* left atrial appendage in patients with atrial fibrillation or flutter not addressed by resection or exclusion at a time of the implant
* hemodynamically significant or symptomatic carotid artery stenosis prior to low-intensity protocol anticoagulation initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Survival-free rate of thromboembolic and hemorrhagic events | 12 months
  12 month survival-free rate of thromboembolic events (i.e. pump thrombosis, disabling stroke MRS>3) and hemorrhagic events (major bleeding, hemorrhagic stroke).

SECONDARY OUTCOMES:
Adverse Events | 12 months
  Adverse Event rates as assessed per INTERMACS definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Netuka, MD, Ph.D., Principal Investigator — Institute for Clinical and Experimental Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Netuka I, Sood P, Pya Y, Zimpfer D, Krabatsch T, Garbade J, Rao V, Morshuis M, Marasco S, Beyersdorf F, Damme L, Schmitto JD. Fully Magnetically Levitated Left Ventricular Assist System for Treating Advanced HF: A Multicenter Study. J Am Coll Cardiol. 2015 Dec 15;66(23):2579-2589. doi: 10.1016/j.jacc.2015.09.083. PMID 26670056
- [Background] Mehra MR, Naka Y, Uriel N, Goldstein DJ, Cleveland JC Jr, Colombo PC, Walsh MN, Milano CA, Patel CB, Jorde UP, Pagani FD, Aaronson KD, Dean DA, McCants K, Itoh A, Ewald GA, Horstmanshof D, Long JW, Salerno C; MOMENTUM 3 Investigators. A Fully Magnetically Levitated Circulatory Pump for Advanced Heart Failure. N Engl J Med. 2017 Feb 2;376(5):440-450. doi: 10.1056/NEJMoa1610426. Epub 2016 Nov 16. PMID 27959709
- [Background] Netuka I, Kvasnicka T, Kvasnicka J, Hrachovinova I, Ivak P, Marecek F, Bilkova J, Malikova I, Jancova M, Maly J, Sood P, Sundareswaran KS, Connors JM, Mehra MR. Evaluation of von Willebrand factor with a fully magnetically levitated centrifugal continuous-flow left ventricular assist device in advanced heart failure. J Heart Lung Transplant. 2016 Jul;35(7):860-7. doi: 10.1016/j.healun.2016.05.019. Epub 2016 May 31. PMID 27435529
- [Derived] Netuka I, Ivak P, Tucanova Z, Gregor S, Szarszoi O, Sood P, Crandall D, Rimsans J, Connors JM, Mehra MR. Evaluation of low-intensity anti-coagulation with a fully magnetically levitated centrifugal-flow circulatory pump-the MAGENTUM 1 study. J Heart Lung Transplant. 2018 May;37(5):579-586. doi: 10.1016/j.healun.2018.03.002. Epub 2018 Apr 11. PMID 29655662